CLINICAL TRIAL: NCT07234370
Title: Distal Radial Fractures in Adult Patients: 4 Weeks Versus 6 Weeks of Cast Immobilization-A Randomized Controlled Trial
Brief Title: Distal Radial Fractures in Adult Patients: 4 Weeks Versus 6 Weeks of Cast Immobilization
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Mohammad Zeeshan Haider, Resident Doctor, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R.C-LNH-Orthpedics-05/2025/52
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Fracture Forearm; Radius Distal Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Splints; POLR1G protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast immobilization for four weeks (Experimental): Scotch cast immobilization for a period of four weeks applied to distal radius fractures.
  Interventions: Procedure: Short Arm Cast for Distal Radius Fracture for four weeks
- Cast immobilization for six weeks (Active Comparator): Scotch cast immobilization for a period of six weeks applied to distal radius fractures
  Interventions: Procedure: Short Arm Cast for Distal Radius Fracture for six weeks

INTERVENTIONS:
Procedure: Short Arm Cast for Distal Radius Fracture for four weeks — Scotch cast immobilization below elbow for four weeks
  Other Names: Splint; Cast
  Arms: Cast immobilization for four weeks
Procedure: Short Arm Cast for Distal Radius Fracture for six weeks — Scotch cast immobilization below elbow for six weeks
  Other Names: Splint; Cast
  Arms: Cast immobilization for six weeks

SUMMARY:
Post-intervention outcomes comparing casting in distal radius fractures of four weeks versus six weeks.

DETAILED DESCRIPTION:
Cast immobilization for 6 weeks remains the mainstay of therapy for distal radius fractures. To challenge the therapeutic time frame, participants will be randomized into two arms, and the treatment arm will undergo immobilization for 4 weeks. Outcomes will be assessed at cast removal and then at 3 and 6 months prospectively using the Quick-DASH score and the DASH score (only at 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with DRF undergoing conservative management with cast immobilization
* Age between 18 to 50 years.

Exclusion Criteria:

* Any syndromic patients
* Any patients with musculoskeletal disease
* Patients having osteoporosis
* Post-menopausal females
* Smokers
* Ages less than 18 or greater than 50
* Patients presenting with intra-articular fractures

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Quick Disability of Arm, Shoulder, and Hand Score (Quick DASH) | Four weeks (Cast Removal)
  Quick Disability of Arm, Shoulder, and Hand (Quick DASH) score is calculated using a formula based on responses to an 11-item questionnaire. Scores range from 0 to 100, where 0 indicates no disability and 100 indicates the most severe disability.
Quick Disability of Arm, Shoulder, and Hand (Quick DASH) | Six weeks (Cast Removal)
  Quick Disability of Arm, Shoulder, and Hand (Quick DASH) score is calculated using a formula based on responses to an 11-item questionnaire. Scores range from 0 to 100, where 0 indicates no disability and 100 indicates the most severe disability.
Quick Disability of Arm, Shoulder, and Hand (Quick DASH) | 3 months after cast removal
  Quick Disability of Arm, Shoulder, and Hand (Quick DASH) score is calculated using a formula based on responses to an 11-item questionnaire. Scores range from 0 to 100, where 0 indicates no disability and 100 indicates the most severe disability.
Quick Disability of Arm, Shoulder, and Hand (Quick DASH) | 6 months after cast removal
  Quick Disability of Arm, Shoulder, and Hand (Quick DASH) score is calculated using a formula based on responses to an 11-item questionnaire. Scores range from 0 to 100, where 0 indicates no disability and 100 indicates the most severe disability.
Disability of Arm, Shoulder, and Hand Score | 6 months post-removal of cast immobilizations
  The Disability of Arm, Shoulder, and Hand Score (DASH) is a 30-item questionnaire with scores ranging from 1 to 5 for each item. The final scores are formulated from 0 to 100, where a higher score indicates greater disability and a lower score indicates little to no disability.

SECONDARY OUTCOMES:
Radial Deviation | 6 months post-cast immobilization removal
  Radial deviation ranges from 15-25°. More deviation suggests more joint movement and is associated with better outcomes.
Ulnar Deviation | 6 months post-cast immobilization removal.
  Ulnar deviation ranges from 30-45 °. More deviation suggests more joint movement and is associated with better outcomes.
Dorsiflexion | 6 months post-cast immobilization removal.
  Dorsiflexion ranges from 8-26 °. More flexion suggests more joint movement and is associated with better outcomes.
Palmar Flexion | 6 months post-cast immobilization removal.
  Palmar flexion ranges from 70-90 °. More flexion suggests more joint movement and is associated with better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nabeel Aamir Syed, MBBS, MD, Principal Investigator
Locations (1):
- Liaquat National Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No